CLINICAL TRIAL: NCT05291975
Title: Clinical Efficacy and Human Factors Validation Testing for Prescription Home Use of the Erchonia Corporation EVRL™ for Providing Temporary Relief of Diabetic Peripheral Neuropathy Foot Pain
Brief Title: Clinical Efficacy and Human Factors Validation Testing of the Erchonia EVRL for Providing Temporary Relief of Diabetic Peripheral Neuropathy Foot Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-DPN-HOME
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Neuropathy, Diabetic; Neuropathy;Peripheral; Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies; Neuritis; Neuropathy, Painful

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Erchonia® EVRL™ (Active Comparator): The Erchonia® EVRL™ is made up of (1) 635 nanometers red laser diode and (1) 405 nanometers violet laser diode mounted in a portable handheld device.
  Interventions: Device: Erchonia® EVRL™
- Placebo Laser (Placebo Comparator): The Placebo Laser has the same appearance as the Erchonia® EVRL™ but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia® EVRL™ — The Erchonia® EVRL™ is made up of (1) 635 nanometers red laser diode and (1) 405 nanometers violet laser diode mounted in a portable handheld device. The diodes are positioned approximately 3 to 6 inches from the top of the foot. The treatments will be self-administered by the subject at his or her's place of residence, two times per day for 21 days. Each procedure administration lasts 5 minutes per foot, for a total of 10 minutes.
  Arms: Erchonia® EVRL™
Device: Placebo Laser — The Placebo Laser has the same appearance as the Erchonia® EVRL™ but does not emit any therapeutic light. The diodes are positioned approximately 3 to 6 inches from the top of the foot. The treatments will be self-administered by the subject at his or her's place of residence, two times per day for 21 days. Each procedure administration lasts 5 minutes per foot, for a total of 10 minutes.
  Arms: Placebo Laser

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® EVRL™, manufactured by Erchonia Corporation (the Company), in providing prescription home use application for temporary relief of diabetic neuropathy foot pain in individuals diagnosed with diabetic neuropathy by a suitably qualified and licensed health professional.

DETAILED DESCRIPTION:
Human Factors Validation Testing will initially be conducted to valuate a lay person's ability to understand and apply as applicable the information contained in the EVRL™ Use Device Proper Use Reference Guide, and device packaging and labeling materials to correctly, safely, and successfully activate and operate the EVRL™ to administer the treatment; and to identify any and all use difficulties, problems and errors, including those pertaining to critical tasks and close calls demonstrated by the lay person during device operation, and to subsequently mitigate each identified instance of use error through device and/or materials modification, and to subsequently evaluate the effectiveness of each modification, as applicable

Phase Two will commence following the successful completion of Phase One. Phase Two comprises the performance of a double-blind, randomized, placebo-controlled, clinical study of the efficacy of the Erchonia® EVRL™, manufactured by Erchonia Corporation (the Sponsor), for prescription home use application in providing temporary relief of diabetic peripheral neuropathy foot pain.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with diabetes induced peripheral neuropathy by a suitably qualified and licensed health professional within the past 6 months
* Over the age of 18 years of age
* Able to read and write English.
* Constant feet pain on-going over at least the past 3 months.
* If using analgesics (pain medication), you must be on a stable analgesic regimen (i.e., no changes to the prescribed analgesic regimen) over a period of at least 14 days prior to enrollment; and willing and able to not have planned upward dose titration of analgesics during the study period. You may elect to decrease analgesic use during the study. Cannabis prescribed for medicinal purposes would qualify as an analgesic in this context.
* Willing and able to refrain from engaging in any non-study procedure therapies for the management of foot pain throughout the course of study participation, including conventional therapies such as physical therapy, occupational therapy and hot or cold packs, as well as alternative therapies such as chiropractic care and acupuncture.
* Agrees to refrain from taking a dosage of analgesic (pain medication) for at least 6 hours before a scheduled VAS foot pain rating is to be recorded.
* Subjects' degree of foot pain on the 0-100 VAS, with "0" being no pain and "100" being worst pain imaginable, is 50 or greater.

Exclusion Criteria:

* Pregnant or think you might be pregnant.
* Open wounds (sores, cuts, ulcers, etc) around the feet
* Cancerous growths around the feet
* Difficulty with hand dexterity sufficient to impact ability to administer treatments with the laser such as from severe arthritis in the hands, Multiple Sclerosis, Cerebral Palsy, Parkinson's Disease, Huntington's Disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - CiC Foot & Ankle, Phoenix, Arizona
  - Laser Chiropractic, West Covina, California
  - Cesar A. Lara M.D. Weight Loss & Wellness, Dunedin, Florida
  - FRANCO & CO Podiatric Medicine & Surgery, Miramar, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia® EVRL™ | Placebo Laser
Started | 33 | 31
Completed | 33 | 27
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia® EVRL™ | Placebo Laser | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.39 (8.35) | 64.74 (9.08) | 66.10 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 18 | 16 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19 | 17 | 36
  Hispanic | 8 | 7 | 15
  African American | 2 | 6 | 8
  Asian / Pacific Islander | 1 | 1 | 2
  Other | 3 | 0 | 3
Duration Since Onset of Foot Pain [Mean (Standard Deviation); unit: months] — The duration since onset of foot pain is recorded in months
  months | 93.33 (89.94) | 79.52 (97.63) | 86.64 (92.52)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 30% or Greater Change in Pain Rating on the Visual Analog Scale (VAS)
Description: The Visual Analog Scale (VAS) from baseline to endpoint (6 weeks) measurement is calculated for each subject. Individual subject success is defined as a 30% or greater change in VAS pain scores across the evaluation period. A negative (-) percent change indicates a decrease in pain level and is positive for individual subject success. A lower Visual Analog Scale pain score from baseline to study endpoint represents a better outcome, whereas a higher score from baseline to study endpoint represents a worse outcome.
  For the primary study outcome, the overall study success is defined as a 35% or greater difference between the proportion (number) of individual successes in each treatment group.
Time Frame: Baseline and 3 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia® EVRL™ | Placebo Laser
Number analyzed (Participants) | 33 | 31
participants | 24 | 9

2. Secondary Outcome: Satisfaction With Study Outcome
Description: At treatment endpoint, the subject was asked to rate how satisfied he or she was with any overall change in foot pain attained following the procedure administration phase with the Erchonia EVRL Laser, using the following five-point scale:
  Very Satisfied Somewhat Satisfied Neither Satisfied nor Dissatisfied Not Very Satisfied Not at All Satisfied
  Results are reported as the number of subjects who reported being 'Very Satisfied' or 'Somewhat Satisfied' with the study outcome.
Time Frame: Baseline and 3 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia® EVRL™ | Placebo Laser
Number analyzed (Participants) | 33 | 31
participants | 20 | 8

3. Secondary Outcome: Four Weeks Post Procedure Change in Foot Pain Visual Analog Scale (VAS) Score
Description: The VAS is a straight line scale that is marked on one end with a '0' for 'no pain' and at the other end with '100' for 'worse pain imaginable.' A higher score on the VAS indicates a greater level of pain, and a lower score indicates a lower level of pain.A decrease in the VAS pain rating indicates a reduction in foot pain and is positive for study success. An increase in the VAS pain rating indicates a worsening of foot pain and is negative for study success. The mean change in foot pain score recorded on the Visual Analog Scale (VAS) from baseline to 4 weeks post treatment was calculated for each treatment group.
Time Frame: Baseline and 7 Weeks
Population: Five (5) participants in the active group and seven (7) participants in the placebo group did not return for the four (4)-week post-procedure follow-up visit. These participants were recorded as "Lost to Follow-up."
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erchonia® EVRL™ | Placebo Laser
Number analyzed (Participants) | 28 | 24
units on a scale | -34.32 (33.61) | -13.41 (28.07)

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Erchonia® EVRL™ | Placebo Laser
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT05291975/Prot_SAP_ICF_000.pdf